CLINICAL TRIAL: NCT01494870
Title: Management of Acute Myocardial Infarction in the Presence of Left Bundle Branch Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samara Regional Cardiology Dispensary (Other)
Responsible Party: Principal Investigator, Ass.Prof. Dmitry Duplyakov M.D., Ph.D., Medical Director, Cardiology Department, Samara Regional Cardiology Dispensary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOKKD-01
Record Dates: First submitted 2011-12-13; First posted 2011-12-19 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; percutaneous coronary intervention; left bundle branch block
MeSH Terms: conditions — Acute Coronary Syndrome; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PCI — urgent PCI on admission

SUMMARY:
The primary objective of this study is to propose new treatment algorithm (strategy) for patients with Acute Coronary Syndrome (ACS) and left bundle-branch block (LBBB).

DETAILED DESCRIPTION:
Current recommendations on the treatment of acute coronary syndrome (ACS) dictate urgent reperfusion therapy in the case of evolving myocardial infarction with ST-segment elevation (STEMI). Optimal use of PCI (preferably) or thrombolysis in this situation requires a rapid and correct diagnosis.

According to the ESC'2008 and ACC/AHA'2009 focused update guidelines patients admitted to the hospital within 12 hours after the onset of chest pain with new (or presumably new) left bundle-branch block (LBBB) should be treated like patients having STEMI (class I, level A). However, it is well-known that in patients with concomitant LBBB, the ECG manifestations of acute myocardial injury may be masked.

ACS may occur in a patient with "true old" LBBB (when doctor has/has not an ability to compare the new ECG with the previous one) or (presumably) new LBBB.

There is a high risk of non receiving appropriate therapy or of receiving inappropriate therapy (thrombolysis instead of LMWH/UFH/fondaparinux).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* Ischemic discomfort (ie, ischemic chest pain or equivalent) at rest ≥20 minutes within previous 24 hours.
* Any (new, presumably new, or old) LBBB on the prehospital (ambulance) or admission ECG.
* Urgent coronary angiography (followed, when indicated, by PCI), ideally within 90 minutes after admission

Exclusion Criteria:

* all-comers design

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
mortality | 30 days

SECONDARY OUTCOMES:
Number of participants survived | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Samara Regional Cardiology Dispansery, Samara, Russia